CLINICAL TRIAL: NCT05275920
Title: Building Electronic Tools To Enhance and Reinforce CArdiovascular REcommendations - Heart Failure (BETTER CARE-HF)
Acronym: BETTER CARE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-00644
Record Dates: First submitted 2022-02-09; First posted 2022-03-11 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Best Practice Alert [BPA]; In-Basket message; Mineralocorticoid Receptor Antagonists [MRA]; guideline-directed medical therapy [GDMT]; Clinical decision support
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Best Practice Alert group (Experimental): Providers will receive a BPA at the time of visit for patients with HFrEF who are not on MRA (and who do not have contraindication to MRA). This alert will display the patient's current HFrEF therapies, EF, blood pressure, potassium, and glomerular filtration rate. The alert will give access to an outpatient heart failure order set, and also provide links to the most recent guidelines.
  Interventions: Other: Best Practice Alert (BPA)
- In-Basket Message group (Experimental): Providers will receive a monthly in-basket messages linking to a list of patients who have been seen in the past 2 months or will be seen in the upcoming month with HFrEF who are not on MRA (and who do not have contraindication to MRA). This list will display each patient's current hFrEF therapies, EF, blood pressure, potassium, glomerular filtration rate, date of last visit, and date of next visit. From the list, providers can access the patient's chart, order medications, and document communication with the patient.
  Interventions: Other: In-Basket Message
- Control group (No Intervention): Patients who will receive the current standard practice of care (no BPA or in-basket message)

INTERVENTIONS:
Other: Best Practice Alert (BPA) — A BPA will fire in the EHR reminding care providers of the best practice when prescribing medical therapies for heart failure patients.
  Arms: Best Practice Alert group
Other: In-Basket Message — An In-Basket message will be sent biweekly to care providers with a reminder of the best practice when prescribing medical therapies for heart failure
  Arms: In-Basket Message group

SUMMARY:
Building Electronic Tools To Enhance and Reinforce CArdiovascular REcommendations - Heart Failure (BETTER CARE-HF) is a pragmatic, cluster-randomized, three-arm intervention trial that will compare the effectiveness of two targeted clinical decision support (CDS) intervention tools (best practice alert (BPA) and automated in-basket massage) to inform providers when a patient with heart failure and reduce ejection fraction (HFrEF) is not on appropriate medical therapy, as compared to usual care.

DETAILED DESCRIPTION:
An estimated 68,000 deaths per year nationwide can be attributed to gaps in care for patients with heart failure and reduced ejection fraction (HFrEF), with the majority being due to lack of mineralocorticoid receptor antagonists (MRA). Despite proven benefits in randomized trials, class I guideline recommendations, and published clinical performance measures, patients with HFrEF are often not on guideline-directed medical therapy (GDMT). While successful interventions for improvement in prescription of GDMT have often included multidisciplinary approaches with dedicated staff, the relatively high cost of hiring additional personnel has led to an interest in electronic health record (EHR)-based interventions. Prior studies on EHR-based interventions in this arena have mainly been conducted in the inpatient setting, which is limited to one encounter during acute hospitalization, a setting often complicated by renal dysfunction or hypotension that can limit prescription of MRA. The development and study of outpatient EHR-based alerts for HFrEF GDMT are needed. Two types of outpatient EHR-based interventions include best practice alerts (BPA) and automated in-basket messages. Both of these methods have limited data, with some studies showing benefit and others demonstrating provider fatigue and burnout. To our knowledge, there is no study that has directly compared these different types of EHR-based interventions.

BETTER CARE - HF is a pragmatic, cluster-randomized, three-arm intervention trail that will compare the effectiveness of two targeted CDS intervention tools (BPA and automated in-basket message) as compared to usual care on the primary outcome of MRA prescription at end of study period.

ELIGIBILITY:
Inclusion Criteria:

* Cardiologist visit
* Transthoracic echocardiogram with the most recent EF >= 40%

Exclusion Criteria:

* Hypotension: SBP < 95
* Hyperkalemia: most recent K > 5.1, or any K >5.5
* Renal dysfunction: eGFR < 30
* Ventricular assist device
* Hospice care
* Cardiac amyloid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2211 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Mukhopadhyay, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Derived] Mukhopadhyay A, Reynolds HR, King WC, Phillips LM, Nagler AR, Szerencsy A, Saxena A, Klapheke N, Katz SD, Horwitz LI, Blecker S. Impact of Visit Volume on the Effectiveness of Electronic Tools to Improve Heart Failure Care. JACC Heart Fail. 2024 Apr;12(4):665-674. doi: 10.1016/j.jchf.2023.11.002. Epub 2023 Nov 15. PMID 38043045
- [Derived] Mukhopadhyay A, Reynolds HR, Phillips LM, Nagler AR, King WC, Szerencsy A, Saxena A, Aminian R, Klapheke N, Horwitz LI, Katz SD, Blecker S. Cluster-Randomized Trial Comparing Ambulatory Decision Support Tools to Improve Heart Failure Care. J Am Coll Cardiol. 2023 Apr 11;81(14):1303-1316. doi: 10.1016/j.jacc.2023.02.005. Epub 2023 Mar 5. PMID 36882134
- [Derived] Mukhopadhyay A, Reynolds HR, Xia Y, Phillips LM, Aminian R, Diah RA, Nagler AR, Szerencsy A, Saxena A, Horwitz LI, Katz SD, Blecker S. Design and pilot implementation for the BETTER CARE-HF trial: A pragmatic cluster-randomized controlled trial comparing two targeted approaches to ambulatory clinical decision support for cardiologists. Am Heart J. 2023 Apr;258:38-48. doi: 10.1016/j.ahj.2022.12.016. Epub 2023 Jan 11. PMID 36640860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Best Practice Alert Group | In-Basket Message Group | Control Group
Started | 755 | 812 | 644
Completed | 755 | 812 | 644
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Practice Alert Group | In-Basket Message Group | Control Group | Total
Number analyzed (Participants) | 755 | 812 | 644 | 2211
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73.0 [64.0 to 81.0] | 73.0 [65.0 to 83.0] | 74.0 [63.0 to 81.0] | 73.0 [64.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 209 | 204 | 633
  Male | 535 | 603 | 440 | 1578
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 103 | 82 | 66 | 251
  Not Hispanic or Latino | 600 | 668 | 532 | 1800
  Unknown or Not Reported | 52 | 62 | 46 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 28 | 28 | 27 | 83
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 4
  Black or African American | 78 | 57 | 56 | 191
  White | 490 | 586 | 448 | 1524
  More than one race | 75 | 75 | 46 | 196
  Unknown or Not Reported | 81 | 66 | 62 | 209
Region of Enrollment [Number; unit: participants]
  United States | 755 | 812 | 644 | 2211

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Prescribed Mineralocorticoid Receptor Antagonists (MRA) During Study
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Alert Group | In-Basket Message Group | Control Group
Number analyzed (Participants) | 755 | 812 | 644
Participants | 224 | 127 | 75

2. Secondary Outcome: Number of Participants Prescribed to Beta-blocker (BB), Angiotensin Converting Enzyme (ACE) Inhibitor, Angiotensin Receptor Blocker (ARB), or Angiotensin Receptor/Neprilysin Inhibitor (ARNI) During Study
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Alert Group | In-Basket Message Group | Control Group
Number analyzed (Participants) | 755 | 812 | 644
Participants | 87 | 94 | 85

ADVERSE EVENTS:
Time Frame: Up to 90 days after intervention completion, an average of 6 months
Description: Assessed using electronic health record (EHR) data.
Groups:
- Best Practice Alert Group - Prescribed MRA: Participants in the Best Practice Alert group who were prescribed MRA.
- In-Basket Message Group - Prescribed MRA: Participants in the In-Basket Message group who were prescribed MRA.
- Control Group - Prescribed MRA: Participants in the control group who were prescribed MRA.
- Best Practice Alert Group - Not Prescribed MRA: Participants in the Best Practice Alert group who were not prescribed MRA.
- In-Basket Message Group - Not Prescribed MRA: Participants in the In-Basket Message group who were not prescribed MRA.
- Control Group - Not Prescribed MRA: Participants in the control group who were not prescribed MRA.
Arm/Group | Best Practice Alert Group - Prescribed MRA | In-Basket Message Group - Prescribed MRA | Control Group - Prescribed MRA | Best Practice Alert Group - Not Prescribed MRA | In-Basket Message Group - Not Prescribed MRA | Control Group - Not Prescribed MRA
All-Cause Mortality (participants affected / at risk) | 2/224 | 0/127 | 0/75 | 0/531 | 5/685 | 5/569
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/127 | 0/75 | 0/531 | 0/685 | 0/569
Other Adverse Events (participants affected / at risk) | 35/224 | 12/127 | 8/75 | 37/531 | 44/685 | 31/569
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Best Practice Alert Group - Prescribed MRA (N=224) | In-Basket Message Group - Prescribed MRA (N=127) | Control Group - Prescribed MRA (N=75) | Best Practice Alert Group - Not Prescribed MRA (N=531) | In-Basket Message Group - Not Prescribed MRA (N=685) | Control Group - Not Prescribed MRA (N=569)
Hyperkalemia (Renal and urinary disorders) | 30 | 12 | 8 | 37 | 43 | 31
Significant Hyperkalemia (Renal and urinary disorders) | 12 | 8 | 3 | 14 | 15 | 12
Newly documented adverse reaction/intolerance to MRA (General disorders) | 6 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT05275920/Prot_SAP_000.pdf